CLINICAL TRIAL: NCT04434339
Title: A Comparison Between Ultrasound-guided Erector Spinae Plane Block and Transversus Abdominis Plane Block for Postoperative Analgesia of Adult Patients Undergoing Ovarian Cancer Surgery Under General Anesthesia: Randomized, Controlled Study.
Brief Title: Ultrasound-guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block for Postoperative Analgesia of Adult Patients Undergoing Ovarian Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-104-2020
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain Management
Keywords: erector spinae; block; pain; transversus; abdominis
MeSH Terms: conditions — Bites and Stings; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): "ESP block group" ,Patients received preoperative US guided ESP block on BOTH sides to be operated upon 30 minutes before being transferred to the OR
  Interventions: Procedure: erector spinae block
- group 2 (Experimental): "TAB group" ,Patients received bilateral lower TAB 30 min before being transferred to the OR
  Interventions: Procedure: transversus abdominis block
- group 3 (No Intervention): "the control group", Patients will not receive any block.

INTERVENTIONS:
Procedure: erector spinae block — A volume of 20 ml for each side of erector spinae plane with 0.25% plain bupivacaine
  Other Names: erector spinae plane block
  Arms: group 1
Procedure: transversus abdominis block — A volume of 20 ml for each side of transversus abdominis plane with 0.25% plain bupivacaine
  Other Names: transversus abdominis plane block
  Arms: group 2

SUMMARY:
Postoperative pain is one of the greatest patient concerns following any surgery. Although an increased emphasis has been placed on pain management, approximately 80% of surgical patients report postoperative pain with 86% of patients rating their pain as moderate, severe, or extreme.

In recent years, the increasing adoption of ultrasound-guided regional anesthesia for acute pain management parallels the rapid rise in the availability of ultrasound machines, facilitating description of a number of important fascial plane blocks blocking the dorsal, lateral and anterior cutaneous nerves of the thorax and abdomen. These new descriptions in blocks are supposed to be an advance in regional anesthesia due to its simplicity and lack of complications. These include the transversus abdominis plane block, rectus sheath block, quadratus lumborum block, pectoralis nerve block, serratus plane block, retrolaminar block, and now the Erector spinae block.

Although ESP and TAB blocks successfully reduced postoperative opioid consumption in previous studies, no study has ever compared their efficacy in postoperative analgesia of adult patients undergoing ovarian cancer surgery under general anesthesia thus in this randomized controlled study we are aiming to fill this gap in the literature.

Hypothesis Analgesia provided by the erector spine plane block is superior to that of transversus abdominis block in patients undergoing ovarian cancer surgery under general anesthesia.

DETAILED DESCRIPTION:
Introduction:

Postoperative pain is one of the greatest patient concerns following any surgery. Although an increased emphasis has been placed on pain management, approximately 80% of surgical patients report postoperative pain with 86% of patients rating their pain as moderate, severe, or extreme.

In recent years, the increasing adoption of ultrasound-guided regional anesthesia for acute pain management parallels the rapid rise in the availability of ultrasound machines, facilitating description of a number of important fascial plane blocks blocking the dorsal, lateral and anterior cutaneous nerves of the thorax and abdomen. These new descriptions in blocks are supposed to be an advance in regional anesthesia due to its simplicity and lack of complications. These include the transversus abdominis plane block, rectus sheath block, quadratus lumborum block, pectoralis nerve block, serratus plane block, retrolaminar block, and now the Erector spinae block.

The TAP is a potential anatomical space that lies between transversus abdominis and internal oblique muscles, where local anesthetic can be deposited, creating a non-dermatomal "field block.".This block can be placed before or during a surgery either by ultrasound guidance or by landmarking through the triangle of Petit (inferior lumbar triangle). Blocks can be placed either intra-abdominally prior to abdominal fascial closure or by transdermal injection. Transversus abdominis plane (TAP) blocks can provide reliable relief of somatic incisional pain. However, the lack of reliable visceral pain relief with TAP blocks may necessitate additional modes of analgesia.

Previous studies have investigated the efficacy of TAP blocks in benign gynecology, general surgery,and non-ovarian gynecologic oncology.These studies have had mixed outcomes, but a recent meta-analysis has demonstrated an overall reduction in pain and opioid usage associated with TAP blocks in laparotomy.

Since its first description by Forero et al. there have been many articles and case reports including an increasingly number of indications for the ESP block: chronic and acute pain treatment , rib fractures management in the emergency setting, treatment of abdominal surgical pain , hip arthroplasty , analgesic management in breast surgery,or in spinal surgery.

The ESP block targets the erector spinae plane, which lies between the anterior surface of the cephalon-caudal oriented erector spinae muscles (that arise from and insert into various bony components of the vertebral column, for example, from spinous process to spinous process, rib to rib, and transverse process to transverse process and the posterior surface of the spinal transverse processes. LA is deposited in the fascial plane deep to the erector spinae muscle and superficial to the tips of the transverse processes, from where it diffuses to the dorsal and ventral rami of spinal nerves, achieving an extensive multi-dermatomal sensory block of the posterior, lateral, and anterior thoracic wall .

ESP block could result in both visceral and somatic abdominal analgesia if the injection were performed at a lower thoracic level.as the local anesthetic penetrates anteriorly through the intertransverse connective tissue and enters the thoracic paravertebral space where it can potentially block not only the ventral and dorsal rami of spinal nerves but also the rami communicants that transmit sympathetic fibers.

For 2019 about 22,530 women will receive a new diagnosis of ovarian cancer and about 13,980 women will die from ovarian cancer as for The American Cancer Society estimation for ovarian cancer in the United States. oncologic ovarian cancer surgeries performed by general anesthesia (GA),cannot provide adequate postoperative pain control as cytoreductive and staging procedures often involve considerable visceral disruption and incisions above the umbilicus have accessory innervation. and the routine use of parenteral opioids aggravates postoperative sedation, nausea, emesis, impaired oxygenation and depressed ventilation.

Although ESP and TAB blocks successfully reduced postoperative opioid consumption in previous studies, no study has ever compared their efficacy in postoperative analgesia of adult patients undergoing ovarian cancer surgery under general anesthesia thus in this randomized controlled study we are aiming to fill this gap in the literature.

Aim of the work Aims to evaluate the analgesic effects of combined general with ultrasound-guided erector spinae block versus that of combined general with transversus abdominis block in patients undergoing major ovarian cancer surgery 1. Inclusion criteria female Patients undergoing ovarian cancer surgery under general anesthesia with ASA I-II and Age ≥ 18 and ≤ 65 Years 2. Exclusion criteria

* Patient refusal.
* uncooperative patients
* Cardiovascular disease in the form of Uncontrolled hypertension, IHD, AF, cardiomyopathy with EF <50%
* Cerebrovascular insufficiency in the form of TIAs, REND, stroke, cerebral hemorrhage, brain tumour, epilepsy
* Coagulation defects with INR>1.5 platelets count< 80000
* hepatic insufficiency with ALT and AST > twice normal, total bilirubin >1.5 , PC < 80%.
* Hypersensitivity to the study drugs.
* Pregnant patients
* patients receiving vasoactive drugs or beta blockers V. Study Procedures

  1. Randomization (in RCT only) Computer generated sequence will be used for randomization.
  2. Study Protocol After approval of the Research Ethics Committee and written informed consent from all patients, A randomized, prospective, comparative, single blinded as the anesthesiologist who will collect data will be blinded for which block was given study to compare between ultrasound-guided erector spinae plane block and transversus abdominis plane block for postoperative analgesia of adult patients undergoing ovarian cancer surgery under general anesthesia with lower midline incision approach will be conducted on A total of 45 Patients that will be randomly allocated by using computer generated random numbers into Group1: (n=15) "ESP block group" ,Patients received preoperative US guided ESP block on BOTH sides to be operated upon 30 minutes before being transferred to the OR, Group 2: (n=15) "TAB group" ,Patients received bilateral lower TAB 30 min before being transferred to the OR and Group 3: (n=15)"the control group", Patients will not receive any block.

The day before surgery, all patients will be instructed to fast for 6-8 hours. On the day of the operation, the patient will arrive to the preparation room 1 hour before operation, to allow time for the block procedure and a minimum of 30 minutes to pass after the block before induction of general anesthesia, an 18 G cannula insertion, a start of IV fluid drip, and premedication with 0.02-0.03 mg/kg intravenous midazolam will be done. All basic monitoring will be applied (ECG/HR/SpO2/NIBP), and baseline values for HR, SPO2, SBP, DBP and MAP will be documented then every 5 minutes till the patient reaches the operating room.

In group 1 a mark will be applied on the required level (T10) identified as 3rd spinous process caudal to that of T7 which located in the middle of a line passing between the lower tips of the scapulae, the midline (spinous processes) and the injection points 3 cm on either sides from midline. While the patient is in a sitting position with support from a member of staff, Preparation of the field with iodine will be made. The ultrasound transducer is placed in a longitudinal parasagittal orientation using the HFL38X linear multi-frequency 6-13 MHz probe of SonoSite M-Turbo of portable ultrasound system anatomical landmarks will be identified including the transverse process at T10 level and the layers of muscles from posterior to anterior: trapezius-erector spinae. After subcutaneous lidocaine 2% injection a 22-G spinal needle will be inserted under ultrasound guidance in plane, aiming towards the transverse process. After a Gentle contact with the transverse process, a volume of 20 ml for each side with 0.25% bupivacaine will be injected in increments with careful repetitive aspiration to avoid intravascular injection targeting to cover dermatomal levels from T8-T12 as minimum.

In group 2 while the patient is lying supine, the probe will be placed perpendicular to the mid-axillary line between the iliac crest and subcostal margin, the 3 abdominal muscle layers were identified, and the transversus abdominis plane was located between the internal oblique and transversus abdominis muscle. Next, 20 mL of 0.25% bupivacaine will be injected in increments with careful repetitive aspiration to avoid intravascular injection, and drug spread in the plane will be observed. The same procedure will be repeated on the other side of the abdomen.

Then the patient will be transferred to the OR. All basic monitoring will be applied (ECG/HR/SpO2/NIBP) while monitoring of end-tidal CO2 will be initiated after induction of anesthesia and values will be recorded for HR, SPO2 ,SBP,DBP ,MAP and ETCO2 every 5 minutes till the end of the surgery then for 30 minutes from time of reaching PACU.

General anesthesia will be induced with 2 mg/kg propofol, 1μg/kg fentanyl and 0.5 mg/kg atracurium to facilitate endotracheal intubation. After intubation the lungs will be mechanically ventilated to maintain the ETCO2 35-40 mmHg. Anesthesia will be maintained with isoflurane keeping the ET concentration of isoflurane 1-2% to maintain the BIS value 40-60. Atracurium besylate top-up doses 0.1mg/kg will be given based on the response to train of four ulnar nerve stimulation. Additional fentanyl dose of 0.5 µg/kg IV for maximum of 3 µg/kg will be given if HR and /or BP increased more than 20% from baseline in response to surgical stimulation and the total dose of fentanyl will be recorded.

The patient's pain will be monitored and documented using the Numerical Rating Score (NRS) for pain at times 0,30 minutes, 1, 2, 4, 6, 8, 10, 12, 18 and 24 hours.(28)The "zero" point of time will be the moment the patient recovered from general anesthesia. Time to first analgesic requirement will be recorded which is the time from the "zero" point till the NRS is 4 or more.

1 g paracetamol IV will be given every 6 hours regardless the NRS value while rescue medication in the form of 50 mg tramadol IV will be given on demand when NRS score is 4 or more with maximum dose of 1 mg /kg every 6 hours and the total consumption of tramadol will be recorded.

Complications in the form of local anesthetic systemic toxicity, failed block, injury to surrounding structures (peritoneum, vessels, dura ,pleura inform of pneumothorax) will be documented

ELIGIBILITY:
Inclusion Criteria:

* female Patients undergoing ovarian cancer surgery under general anesthesia with ASA I-II and Age ≥ 18 and ≤ 65 Years

Exclusion Criteria:

* Patient refusal.
* uncooperative patients
* Cardiovascular disease in the form of Uncontrolled hypertension, IHD, AF, cardiomyopathy with EF <50%
* Cerebrovascular insufficiency in the form of TIAs, REND, stroke, cerebral hemorrhage, brain tumour, epilepsy
* Coagulation defects with INR>1.5 platelets count< 80000
* hepatic insufficiency with ALT and AST > twice normal, total bilirubin >1.5 , PC < 80%.
* Hypersensitivity to the study drugs.
* Pregnant patients
* patients receiving vasoactive drugs or beta blockers

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
postoperative tramadol consumption | within 24 hours after surgery
  postoperative tramadol consumption in mg

CONTACTS AND LOCATIONS:
Locations (1):
- anesthesia department at Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not for sharing

REFERENCES:
- [Background] 25. .Jiří M.,et al. Postoperative Pain Management. Third updated edition.Mladá fronta a. s., Mezi Vodami 2017.1952/9 26. Tulgar S. et tal Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective,randomized, controlled clinical trial. Journal of Clinical Anesthesia .2018; (49):101-106 27. Canakci, E.et al.The Analgesic Efficacy of Transverse Abdominis Plane Block versus Epidural Block after Caesarean Delivery: Which One Is Effective? TAP Block? Epidural Block?." Pain research & management. 2018. 3562701. 28. Rodriguez CS. Pain measurement in the elderly: a review. Pain Manag Nurs 2001;(2):38-46 29. Altıparmak. B.,et tal. Ultrasound-guided erector spinae plane block versus oblique subcostal transversus abdominis plane block for postoperative analgesia of adult patients undergoing laparoscopic cholecystectomy: Randomized, controlled trial Journal of Clinical Anesthesia. 2019;(57):31-36